

BRANY ID # 18-02-365 Version/Date: v5.5, 24-OCT-2023

**TITLE:** Randomized controlled trial assessing transperineal prostate biopsy to reduce infection complications

#### BRANY ID # 18-02-365 VERSION/DATE: v5.5, 24-OCT-2023

Principal Investigator: Jim C. Hu, MD MPH (contact)

525 E 68th Street, Starr 946

New York, NY 10065 Weill Cornell Medicine Telephone 646.962.9600 Fax 646.962.0715

jch9011@med.cornell.edu

Edward M. Schaeffer, MD PhD

NMH/Arkes Family Pavilion Suite 2300

676 N Saint Clair Chicago, IL 60611 Northwestern University Telephone 312.908.8145 <u>e-</u> schaeffer@northwestern.edu

Mohamad Allaf, MD

600 North Wolfe Street, Park 223

Baltimore, MD 21287 Johns Hopkins University Telephone 410.502.7710

Fax 410.502.7711 mallaf@jhmi.edu

rs: Behfar Ehdaie, MD MPH

323 E 68<sup>th</sup> Street New York, NY 10065

Memorial Sloan Kettering Cancer Center

Telephone 646.422.4406 ehdaieb@mskcc.org

Timothy McClure, MD 525 E 68<sup>th</sup> Street, Starr 900 New York, NY 10065 Weill Cornell Medicine Telephone 646.962.9600 tim9047@med.cornell.edu

Anthony Schaeffer, MD 675 N Saint Clair, Ste 20-150 Chicago, IL 60611 Northwestern University ajschaeffer@northwestern.edu Ashley Ross, MD, PhD

# Co-Investigators:

675 N Saint Clair, Ste 20-150 Chicago, IL 60611 Northwestern University Telephone 312.695.8146 ashley.ross@nm.org

Jeffrey Montgomery, MD 1500 E Medical Center Dr SPC 5913 Ann Arbor, MI 48109 University of Michigan Telephone 734.647.8903 montrose@med.umich.edu

Arvin George, MD 1500 E Medical Center Dr, Floor 2 Ann Arbor, MI 48109 University of Michigan Telephone 734.936.7030 arvigeor@med.umich.edu

John Graham, MD 38 6<sup>th</sup> Avenue, 2<sup>nd</sup> Floor Brooklyn, NY 11217 NewYork-Presbyterian Brooklyn Methodist Hospital Telephone 718.230.7788 jng9008@med.cornell.edu

David Green, MD 58-42 Main Street Flushing, NY 11355 NewYork-Presbyterian Queens Telephone 718.303.3720 dag9025@nyp.org

Gerald Wang, MD 56-45 Main Street Flushing, NY 11355 NewYork-Presbyterian Queens Telephone 718.303.3720 gew9003@nyp.org

Serge Ginzburg, MD
1200 Tabor Rd, 3<sup>rd</sup> Floor
Philadelphia, PA 19141
Einstein Urology
Telephone 215.356.4658
ginzburs@einstein.edu
Keith Kowalczyk, MD
3800 Reservoir Road Northwest, 4<sup>th</sup> Floor
Washington, DC 20007

Georgetown University
Telephone 202.295.0580
keith.kowalczyk@medstar.net

Andres Correa 333 Cottman Avenue Philadelphia, PA 19111 Fox Chase Cancer Center Telephone 215.728.6900 andres.correa@fccc.edu

Benjamin Ristau, MD 263 Farmington Avenue Farmington, CT 06030 University of Connecticut Telephone 860.679.4100 beristau@uchc.edu

Jonathan Shoag, MD 11100 Euclid Avenue Cleveland, OH 44106 Case Western University Telephone 216.844.3009 jxs218@case.edu

Statistician:

Andrew Vickers, PhD 485 Lexington Ave New York, NY 10017 Memorial Sloan Kettering Cancer Center Telephone 646.888.8233 vickersa@MSKCC.org Confidentiality

Statement

This document is confidential and is to be distributed for review only to investigators, potential investigators, consultants, study staff, and applicable independent ethics committees or institutional review boards. The contents of this document shall not be disclosed to others without written authorization from the Principal Investigator.

### **Protocol Summary**

Randomized controlled trial assessing transperineal prostate **Full Title:** 

biopsy to reduce infection complications

Clinical Phase:

**Principal Investigator:** Jim C. Hu, M.D., M.P.H.

Sample Size: N = 1.702

**Study Population:** Men who are aged at least 18 years with: history of Grade Group

> 1 or 2 prostate cancer, first diagnosed prior to date of planned biopsy (active surveillance cohort); clinical concern for the presence of prostate cancer as determined by the treating urologist and prior negative prostate biopsy performed ≤36 months prior to date of planned biopsy (prior negative cohort); Men without previous prostate biopsy (first time prostate biopsy)

**Accrual Period:** Approximately 31 months

Study Design: Prospective, randomized trial with 1:1 ratio to either the

transperineal or transrectal biopsy group. Participants will be

assessed for adverse events, pain and discomfort immediately and

7 days post-biopsy.

**Intervention Description:** Transrectal prostate biopsy (TR-Bx) under local anesthesia is

> currently the most commonly used approach to evaluate for the presence of prostate cancer. A limitation of TR-Bx is the need for

biopsy needles to pass through the rectal mucosa on their

trajectory to the prostate, placing men at high risk of an infectious complication. An alternative method for performing prostate biopsy is via a percutaneous transperineal approach. One limitation of transperineal prostate biopsy (TP-Bx) has been the historic need for it to be performed under general or spinal anesthesia in order for patients to tolerate the multiple required needle passes through the perineal skin. Due to recent technical advances TP-Bx may

now be safely performed under local anesthesia.

**Primary Objective:** To compare infection adverse events of TP-Bx vs. TR-Bx

performed under local anesthesia.

**Secondary Objectives:** To compare other adverse events such as bleeding and urinary

retention. To compare detection rates of clinically significant and

insignificant prostate cancer.

**SCHEMA** 



 4.5 Biopsy Procedure
 12

 4.6 Duration of Follow Up
 12

 5. MEASUREMENT OF OUTCOMES
 13

 5.1 Adverse events
 13

 5.2 Pain, Anxiety and Discomfort
 14

| 5.3 Biopsy Pathology | 14 | 4 |
|----------------------------|----|---|
| STATISTICAL CONSIDERATIONS | | |

# 1. Study Objectives

Primary Objective: The primary objective of this study is to compare the incidence and severity of infectious complications between the transperineal and transrectal approaches to prostate biopsy.

Secondary Objectives: Secondary objectives of this study include comparing the incidence of other adverse events, associated pain, and cancer detection rates between the transperineal and transrectal approaches.

#### 2. Background

Approximately one million transrectal prostate biopsies (TR-Bx) are performed annually in the United States. The number of prostate Bx is expected to increase due to the demographic growth of the aging male population. Moreover, 44% of U.S. men undergoing initial biopsy report having a repeat biopsy within five years. Additionally, more than half of men diagnosed with prostate cancer currently opt for active surveillance, which requires serial repeat biopsy to monitor for disease progression. Therefore, biopsy use will only increase with greater adoption of active surveillance and the greater number of aging men. The safety and effectiveness of this common procedure will impact 1 out of 3 U.S. men at least once during their lifetimes when they undergo biopsy.

Due to the need for biopsy needles to pass through the rectal mucosa on their trajectory to the prostate, TR-Bx is associated with a significant risk of infectious complications. The needle travels through the "dirty" rectal mucosa to the "clean" prostate at least 12 times,<sup>4</sup> and fecal flora may seed the vascular prostate gland and bloodstream, leading to infection.<sup>5,6</sup> One systematic review suggests this rate may be as high as 5%.<sup>7</sup> The United States Preventive Services Task Force (USPSTF) Grade C recommendation for PSA screening considered adverse events associated with biopsy among the harms of PSA-based screening.<sup>8</sup> Despite antibiotic prophylaxis, 44% of men experience bacteriuria and 16% experience bacteremia after TR-Bx.<sup>9</sup>

Furthermore, the risk of post-biopsy infection has increased in recent years due to the growing incidence of antibiotic resistance.<sup>10</sup> Nam first reported an alarming four-fold, population-based increase in post-Bx infection hospital admissions from 0.6% in 1996 to 3.6% in 2005 among 75,190 patients.<sup>11</sup> In particular, men with fluoroquinolone-resistant bacteria in the rectum are at increased risk for post-Bx infection and sepsis,<sup>12</sup> which can result in dire complications such as limb gangrene/amputation, endocarditis, meningitis, disseminated intravascular coagulation (DIC) or death.<sup>13–18</sup>

As an alternative to the transrectal approach, prostate biopsy may be performed percutaneously through the perineal skin. Due to avoidance of the rectum, transperineal prostate biopsy (TP-Bx) is associated with an overall lower risk of infectious complications. At some centers, this has obviated the need for perioperative antibiotics, which is reinforced by the Society of Interventional Radiology Guidelines. <sup>19,20</sup> One additional benefit of TP-Bx is that this procedure offers better sampling of the anterior prostate, which is missed with the transrectal approach in men with larger prostate volumes due to benign prostatic hyperplasia. <sup>21</sup> The biopsy core excursion is 2 cm, and therefore sampling of the anterior prostate from the rectum is limited. In contrast, the TP approach has relative ease of access to the anterior prostate. <sup>6</sup> This is reflected

in greater detection of clinically significant prostate cancer in retrospective studies with transperineal<sup>22–25</sup> under general anesthesia (49%-91%) vs. transrectal<sup>24,26–31</sup> Bx approaches (14-42%). Given more than 80% of first-time biopsy nationally are performed without MRItargeting,<sup>32,33</sup> the utility of in-office transperineal vs. transrectal MRI-targeted biopsy must be evaluated as this applies to a large population of men. For instance, the American Urological Association professional guidelines were updated to recommend MRI use for first-time biopsy in early 2020;<sup>34</sup> however, lack of insurance coverage and limited access for urologists to the costly MRI-targeted biopsy platform contribute to a large population of men who need to be evaluated in the repeat biosy setting of active surveillance and prior negative biopsy.

Despite the aforementioned benefits of TP-Bx, this procedure has seen limited adoption due to the historic need for it to be performed under general anesthesia in order for patients to tolerate the required multiple needle sticks to the perineal skin. Additionally, because of the need for biopsy needles to traverse the pelvic floor muscles and vascular prostate apex, TP-Bx is believed to have a higher risk for urinary retention and bleeding as compared to the traditional transrectal approach.

In recent years, the development of novel local anesthetic techniques and needle guides has permitted TP-Bx to be performed in the office setting with a more favorable side-effect profile.<sup>20,35,36</sup> There has, however, been slow adoption of this procedure by only a handful of centers. In fact, national estimates of TP-Bx use place this figure closer to approximately 1-2%.

In this study, we aim to compare the safety, tolerability, and cancer detection rates of TP-Bx versus TR-Bx within the contexts of a randomized clinical trial. The results of this study will provide high level medical evidence regarding which method of prostate biopsy carries the best risk to benefit ratio for men undergoing evaluation for prostate cancer.

### 3. Subject Selection

# 3.1 Study Population

This study will include all men who are recommended to undergo prostate biopsy as part of routine clinical care. Inclusion and exclusion criteria are listed in the following sections.

# 3.2 Inclusion Criteria

- Male sex
- Age ≥18 years
- Active surveillance cohort: History of Grade Group 1 or 2 prostate cancer, first diagnosed prior to date of planned biopsy
- Prior negative cohort: Clinical concern for the presence of prostate cancer as determined by the treating urologist and prior negative prostate biopsy ≤36 months prior to date of planned biopsy
- Men without previous prostate biopsy (first time prostate biopsy)
- Willingness to sign informed consent and adhere to the study protocol

#### 3.3 Exclusion Criteria

- Acute prostatitis within the last 6 months
- PSA > 20 ng/mL in men who have previously undergone prostate biopsy
- Current non-urologic bacterial infection requiring active treatment with antibiotics
- Unfit to undergo prostate biopsy under local anesthesia

- Prior definitive therapy for prostate cancer, such as radiation therapy or partial gland ablation
- Men who have previously undergone prostate biopsy in whom artifact would reduce quality of prostate MRI (extensive orthopedic pelvic metal)
- Contraindication to prostate MRI (claustrophobia, pacemaker, chronic kidney disease) in men who have previously undergone prostate biopsy

## 4. Study Procedures

### 4.1 Study Enrollment and Randomization

Eligible patients will be informed of the study by the study urologist and research staff. Interested participants may also learn more about the study through online resources such as ClinicalTrials.gov or through study informational brochures. All potential subjects will be allowed as much time as needed to consider study participation. Patients choosing to participate in the study will be consented within the privacy of a clinical exam room. Study staff will explain to each potential subject the research objectives, risks and benefits of study participation, and the subjects' rights and responsibilities. For patients who are scheduled for biopsy, electronic consent will also be available via phone. Eligible patients will be contacted by a member of the study team (i.e. investigator or research coordinator), who will explain the study to the patient. The patient will also receive a link to the electronic consent form via email or MyChart message.

This study will utilize either a traditional one-stage or a two-stage consent process. The reason for having the one-stage consent is there are a few sites in which the predominant approach is transperineal. Therefore, this two-stage consent does not work. With the one-stage consent, patients give permission to participate in the study prior to randomization (tradtional RCT consent). With a second-stage consent, subjects who meet all eligibility criteria will sign the firststage consent form. Patients will have the option to sign the consent in person or electronically. First-stage consent will register the subject to the study and will allow investigators to use their data from their medical record and post-biopsy questionnaire responses for research purposes. Subjects who sign first-stage consent will be randomized in a 1:1 ratio to receive TP-Bx or TRBx. The patients' first-stage consent or their traditional one-stage consent will be valid for eight months to accommodate for biopsy scheduling. This will reduce the number of re-consents and align with the standard of care timeline for biopsy procedures. Biopsies are often scheduled as far out eight months from their clinic visit.

Participants will be consented remotely using an electronic version of the informed consent form that follows federal, state, and local regulations, as applicable. We will implement the following procedures for electronic informed consent.

The informed consent document(s) will be sent to the subject or their Legal Authorized Representative (LAR), if applicable, via secure email sent by REDCap prior to the scheduled consent discussion. The subject or LAR will be asked to review the consent document prior and during the consent discussion with a study staff member via phone or approved teleconferencing service (i.e., Zoom). The study staff member will confirm the subject or LAR has read and has the capacity to appreciate all aspects of the information presented in the consent process for the research study. The subject or LAR will be encouraged to ask questions. If agreeing to participate, the subject or LAR will sign the consent form using electronic informed consent (eConsent) via REDCap. A computer, tablet or touch screen phone will be used to capture digital signatures. The person conducting consent will also sign the electronic informed consent (eConsent) document in a contemporaneous manner. Subjects will

be provided with a digital copy of the completed form via email. The informed consent discussion and process will be documented by the study team in the subject's medical record or study record.

If a subject does not have access to a touch screen phone, computer or tablet, cannot work with remote electronic informed consent, or the remote electronic informed consent cannot be obtained for any other reasons, the consent may be conducted and documented at an in-person visit prior to study activities via paper consent form or through REDCap on an ITS tagged device.

The assignment sequence will use randomly permuted blocks of unequal size stratified by urologist, PSA (<4, 4-9.9, ≥10 ng / mL) and biopsy indication (prior negative vs. active surveillance) and implemented by the randomization model in REDCap, which prevents an investigator from learning allocation before a patient is unambiguously registered on study and from changing allocation afterwards, thus ensuring full allocation concealment. For men with prior biopsy, we exclude men with a PSA >20 ng/mL.

For the REDCap randomization model, randomization of subjects will occur on the data collection form where the randomization field is located. Before a subject is randomized, a 'Randomize' button will appear next to that field. When a user (who has been given appropriate 'Randomize' user privileges) clicks that button, a pop-up box will appear that will allow the user to randomize the subject. After a subject has been randomized, the grouping (i.e. transrectal or transperineal biopsy) will become permanently locked and unmodifiable. The randomization field will always be locked and unmodifiable both before and after randomization has occurred for a subject.

Randomization is unblinded, and research coordinators of respective enrolling sites will inform their patients of the assigned cohort.

Subjects randomized to TR-Bx will receive transrectal biopsy. Subjects randomized to TP-Bx will undergo a second consent discussion with the enrolling investigator, where the risks and benefits of transperineal biopsy will be explained. Subjects can then decide whether to undergo standard transrectal biopsy or transperineal biopsy. Subjects who agree to undergo TP-Bx will sign the second-stage consent form.

### 4.2 Data Collection & Confidentiality

Study data will be prospectively collected from patient medical records and patient surveys. In all participating centers, the site-specific research coordinator will perform baseline data acquisition and medical record abstraction. This data will be entered into standardized clinical report forms housed within a REDCap environment and hosted by WCM. Each patient will be assigned a unique study identifier.

REDCap (Research Electronic Data Capture) is a secure, web-based application designed exclusively to support data capture for research studies. The REDCap platform will be partitioned to permit read/write access only to site-specific records such that individual sites will be able to access records for their own subjects, exclusively. REDCap has a secure email and web-based data collection interface that may be utilized for collecting data. The site-specific research coordinator will determine individual patients' preferred method of survey response

and may collect survey data either through mail, telephone, REDCap, or during an in-person visit.

Only the WCM research coordinator will be able to review de-identified data across sites to conduct data quality checks and share data quality with the study biostatistician.

To ensure accuracy of data entered in the REDCap database from source documents (including surveys and medical record abstract), sites will perform 100% visual review and conduct double data entry for a sample (i.e., 10%) of the data.

Data quality checks will be conducted every 6 months, coinciding with Data Safety and Monitoring reviews.

For protocol deviations fitting immediately reportable criteria, the DSMC's primary concern lies with whether the deviation has the potential to negatively impact subject safety or integrity of study data or whether the deviation places subjects at greater risk of harm (including physical, psychological, economic or social harm). If the DSMC makes determinations that the reported protocol deviation impacts either, it may recommend modifications, suspension or termination of the study.

Interim study findings will be communicated in cases where modifications are recommended. The DSMC will require the PI to submit confirmation to the DSMC that the modification(s) have been made, or to submit a reason why the PI did not agree with the DSMC's recommendation.

## 4.3 Study Calendar

| | Month -8 to Day<br>0 | Day 0 | Day 5 to 9 |
|---|---|---|---|
| Eligibility | Xa | | |
| Informed consent | Х | | |
| Demographics | Х | | |
| Medical history <sup>b</sup> | Х | | |
| Physical exam <sup>c</sup> | Х | | |
| Randomization | X | | |
| PSA | Х | | |
| Rectal swab <sup>d</sup> | X | | |
| Prostate Biopsy | | X | |
| Assessment of Adverse Eventse | | | X |
| Concomitant Medications <sup>f</sup> | | X | Х |

<sup>a</sup>To be performed prior to informed consent. <sup>b</sup>Medical comorbidities, indication for biopsy, multiparametric MRI findings, and history of prior biopsy or infection. <sup>c</sup>Height and weight. <sup>d</sup>for transrectal biopsy only.

<sup>e</sup>Assessed by patient questionnaire. Events will be grading using Common Terminology Criteria for Adverse Events (CTCAE) v5.0. <sup>f</sup>Assessed by patient quaestionnaires.

## 4.4 Antibiotic Administration

For patients undergoing a TR-Bx, antibiotic prophylaxis will be administered in accordance with guidelines from the American Urological Association (AUA).<sup>37</sup> No antibiotic prophylaxis will be administered for patients undergoing a TP-Bx.

## 4.5 Biopsy Procedure

A meeting of study investigators will take place before recruitment to review and ensure standardization of biopsies approaches. Investigators will follow the technique described by Kubo et al. to administer lidocaine during TP-Bx.<sup>20</sup> For both transperineal and transrectal approaches, 20 mL of 1% lidocaine will be used, respectively, to standardize local anesthesia. At each site, however, the choice of commercial MRI-targeted biopsy platform will be left to the physicians' discretion.

In both transperineal and transrectal biopsy arms for MRI-targeted biopsy, the number of systematic biopsy cores will be standardized to 12 cores. The technique for TR-Bx is performed as described by Kasivisvanathan et al.<sup>22</sup> A total of 12 systematic biopsy cores will be obtained from the peripheral zone of the prostate at the base, mid gland, and apex. Locations of the 12 systematic cores are: Right lateral base, Right lateral midgland, Right lateral apex, Right medial base, Right medial midgland, Right medial apex, Left lateral base, Left lateral midgland, Left lateral apex, Left medial base, Left medial midgland, and Left medial apex. The technique for TPBx is performed as described by Urkmez et al.<sup>38</sup>. Locations of the systematic cores will be obtained as follows: 2 cores each at Right posterior lateral, Right posterior medial, Left posterior lateral, and Left anterior lateral, and Left anterior lateral, and Left anterior lateral, and Left anterior medial.

In both transperineal and transrectal biopsy arms, the number of targeted biopsy cores will be standardized to 3 cores per target, with a maximum of three ROIs permitted to be chosen for targeted biopsy. MRI-targeted biopsy registration (i.e., matching of the image of the target on MRI with the real-time image of the prostate during biopsy) may be performed by means of visual registration or software-assisted registration.

De-identified video capture of each site's first 10 TP-Bx and TR-Bx will be distributed for review among investigators to monitor for variation in biopsy technique. Deviations from the technique that may occur during routine clinical care will be recorded for each case, monitored by the WCM DSMC and compared between groups. Research coordinators at each site will randomly select 3 TP-Bx and 3 TR-Bx for video upload every 3 months. Investigators will review and discuss during quarterly video-conferences to ensure consistent procedural fidelity throughout the study.

#### 4.6 Duration of Follow Up

Patients will be followed for approximately 7 days following biopsy to evaluate for adverse events. Subjects experiencing an adverse event beyond 7 days stabilization will be followed until resolution or stabilization.

#### 5. Measurement of Outcomes

## 5.1 Adverse events

The primary objective of this study is to compare the incidence and severity of infectious complications experienced by patients undergoing TP-Bx versus TR-Bx. Patients will be assessed for complications by way of electronic questionnaire administered 7±2 days post biopsy using a REDCap site hosted at Weill Cornell Medical Center. For patients unable to complete the questionnaire electronically, responses will be obtained via telephone interview. Any patient indicating that they experienced an adverse event will be contacted by the study team to seek further details. Additionally, all relevant medical records will be requested. Adverse events will be classified in accordance with Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

The primary outcomes are infection rates of TP-Bx versus TR-Bx.

The secondary outcomes are patient-reported pain and anxiety, and comparison of noninfectious complications such as bleeding and urinary retention rates, and cancer detection.

| Timing for assessment of study variables. | | | |
|---|---|---|---|
| Assessment | Baseline<br>Pre-Bx | Day<br>of Bx | 7-days<br>Post-Bx |
| Baseline history and physical exam, screening, consent | ✓ | | |
| Prior Bx (Y/N) | ✓ | | |
| Prior Bx infection (Y/N) | ✓ | | |
| PSA | ✓ | | |
| Indication for Bx | ✓ | | |
| MpMRI findings | ✓ | | |
| Randomization: TR-Bx vs. TP-Bx | ✓ | | |
| Bx infection risk determination for TR-Bx prophylaxis | ✓ | | |
| Bx completed (Y/N) | | ✓ | |
| Bx duration (minutes) | | ✓ | |
| Pain (VAS) | | ✓ | ✓ |
| Discomfort (VAS) | | ✓ | ✓ |
| TMI Anxiety (Likert 5 levels) | | ✓ | |
| Decision regret | | | ✓ |
| Adverse events (Y/N) and Bother UTI | | | J |
| Sepsis | | | ✓ |
| Urinary retention | | | ✓ |

| Fever | ✓ |
|------------------------------------|----------|
| Hematuria | ✓ |
| Hematochezia | ✓ |
| Hematospermia | <b>√</b> |
| UTI diagnosed by HCP | ✓ |
| Unplanned HCP contact | ✓ |
| Qualitative responses | ✓ |
| Bx pathologic outcomes, if cancer: | ✓ |
| Gleason grade group(s) | ✓ |
| Number of cores positive | ✓ |
| Number of cores negative | ✓ |
| Maximum cancer core length | ✓ |
| Targeted Bx positive (Y/N/NA) | ✓ |
| Systematic Bx positive (Y/N) | ✓ |
| Location of positive cores | ✓ |

# 5.2 Pain, Anxiety and Discomfort

A questionnaire will be given to patients immediately after the biopsy and at 7±2 days post-biopsy (Appendix). The questionnaire captures discomfort and pain and fear-anxiety using a numerical rating scale (0-10), with higher scores indicating greater intensity of symptoms. The questionnaire also asks about the presence or absence of adverse events, with reporting of significant adverse events (fever, chills, urinary retention, urinary tract infection, treatment from a doctor) subject to follow-up from study staff.

Infectious complications will be captured as: (1) uncomplicated urinary tract infection (UTI): dysuria, urgency, frequency or hematuria without fever and with or without pyuria (>5 white blood cells per high-powered field or positive leukocyte esterase on urine dipstick) or bacteriuria (≥ 105 colony-forming units/mL); (2) complicated UTI: fever, flank pain, nausea or vomiting with or without pyuria and bacteriuria; (3) urosepsis: criteria for sepsis, severe sepsis, and septic shock<sup>39</sup> were combined and categorized as urosepsis.<sup>40</sup>

# 5.3 Biopsy Pathology

The proportion of men diagnosed with clinically significant cancer and clinically insignificant cancer will be compared by biopsy approach. Detection of prostate cancer will be captured from the final pathology report. We will record the prostate cancer grade, number and location of positive biopsies for transrectal (location: left vs. right, medial vs. lateral, apex, mid, and base) and for transperineal (location: posterior medial, posterior lateral, and anterior), as well as the maximum cancer core length (in mm), and total number of negative cores. In order to compare outcomes, prostate cancer grade will be categorized into insignificant (Gleason grade group 1) and clinically significant (grade group  $\geq 2$ ).<sup>22</sup>

#### 6. Statistical Considerations

We define <u>infection complication</u> as any of the following: (1) fever requiring medical advice or intervention; (2) chills requiring medical advice or intervention; or (3) UTI diagnosed by healthcare professional. We aim to enroll 1,702 (n=682 active surveillance, n=620 prior negative biopsy, n=400 first time biopsy) subjects in this study, with equal randomization between groups. We assume that the infection rate in the transperineal group is 0.5%. Given a one-sided  $\alpha$  of 0.10, the power to reject the null hypothesis of no difference in infection rates will be >80% if the event rate in the transrectal group is 2.0%. The event estimate is consistent with published post-transrectal biopsy infection rates range from 1% to 17.5% and the 2017 AUA prostate biopsy guidelines cite an infection risk of 5-7%. The event estimate is consistent with published post-transrectal biopsy guidelines cite an infection risk of 5-7%.

Analysis of infection, detection of clinically significant cancer (i.e. Grade Group 2+), over-detection of clinically insignificant cancer (i.e. Grade Group 1), presence vs. absence of other biopsy related complication grade 2 or above and, separately, Grade 1 (patient-reported hematuria, hematospermia or hematochezia) will be by logistic regression with site and prior negative vs. active surveillance as fixed effect covariates. The Barnard's test will be used to analyze the data. Absolute risk differences will be calculated by applying the odds ratio from the regression to the prevalence in the transrectal group, with 95% CI obtained by bootstrapping. As a sensitivity analysis for high-grade cancers missed on biopsy, we will include as an event any detection of grade group ≥2 cancer up to two years after randomization, whether detected by subsequent biopsy or upgrading on surgical pathology, as a binary variable. We will also explore whether the relative effects of transperineal biopsy on cancer detection varies by race or diagnostic setting (active surveillance vs. prior negative) by adding race (African ancestry yes or no) or setting (active surveillance vs. prior negative) and the associated interaction terms in two separate logistic regression models.

Rates of missing data are expected to be extremely low because all outcomes are assessed within a short period of time after biopsy. Hence, we do not anticipate having to use statistical methods to handle missing data. However, if rates of missing data are more than 5%, we will implement multiple imputation using chained equations.

To compare the detection of clinically significant cancer biopsy with systematic vs. MRI-targeted biopsy, stratified by transperineal vs. transrectal, the analyses will be conducted separately for the prior negative biopsy and active surveillance cohorts separately. For the prior negative biopsy patients, we will create a model with the outcome of clinically significant cancer and predictors of the linear predictor from the standard Prostate Biopsy Collaborative Group model plus PI-RADS version 2 MRI score and MRI prostate volume. For the active surveillance cohort, we will use a similar approach but use the Canary "base" model for biopsy outcome in active surveillance patients. We will report the increase in discrimination associated with using MRI volume and PIRADS score and conduct decision curve analysis, a decision-analytic technique that weighs the value of avoiding unnecessary biopsy compared to missing high-grade cancer, to assess the clinical utility of the models. Second conduct decision curve analysis and conduct decision curve analysis and conduct decision curve analysis and conduct decision curve analysis and conduct decision curve analysis and conduct decision curve analysis.

#### References

- 1. Loeb S, Carter HB, Berndt SI, Ricker W, Schaeffer EM. Complications after prostate biopsy: data from SEER-Medicare. *J Urol*. 2011;186(5):1830-1834. doi:10.1016/j.juro.2011.06.057
- 2. Welch HG, Fisher ES, Gottlieb DJ, Barry MJ. Detection of prostate cancer via biopsy in the Medicare-SEER population during the PSA era. *J Natl Cancer Inst*. 2007;99(18):1395-1400. doi:10.1093/jnci/djm119
- 3. Cooperberg MR, Carroll PR. Trends in Management for Patients With Localized Prostate Cancer, 1990-2013. *JAMA*. 2015;314(1):80-82. doi:10.1001/jama.2015.6036
- 4. Litwin MS, Tan H-J. The diagnosis and treatment of prostate cancer: A review. *JAMA*. 2017;317(24):2532-2542. doi:10.1001/jama.2017.7248
- 5. Williamson DA, Barrett LK, Rogers BA, Freeman JT, Hadway P, Paterson DL. Infectious complications following transrectal ultrasound-guided prostate biopsy: new challenges in the era of multidrug-resistant Escherichia coli. *Clin Infect Dis.* 2013;57(2):267-274. doi:10.1093/cid/cit193
- 6. Chang DTS, Challacombe B, Lawrentschuk N. Transperineal biopsy of the prostate--is this the future? *Nat Rev Urol.* 2013;10(12):690-702. doi:10.1038/nrurol.2013.195
- 7. Borghesi M, Ahmed H, Nam R, et al. Complications After Systematic, Random, and Image-guided Prostate Biopsy. *Eur Urol.* 2017;71(3):353-365. doi:10.1016/j.eururo.2016.08.004
- 8. US Preventive Services Task Force, Grossman DC, Curry SJ, et al. Screening for prostate cancer: US preventive services task force recommendation statement. *JAMA*. 2018;319(18):1901-1913. doi:10.1001/jama.2018.3710
- 9. Lindert KA, Kabalin JN, Terris MK. Bacteremia and bacteriuria after transrectal ultrasound guided prostate biopsy. *J Urol*. 2000;164(1):76-80. doi:10.1016/S00225347(05)67453-8
- 10. Mosharafa AA, Torky MH, El Said WM, Meshref A. Rising incidence of acute prostatitis following prostate biopsy: fluoroquinolone resistance and exposure is a significant risk factor. *Urology*. 2011;78(3):511-514. doi:10.1016/j.urology.2011.04.064
- 11. Nam RK, Saskin R, Lee Y, et al. Increasing hospital admission rates for urological complications after transrectal ultrasound guided prostate biopsy. *J Urol*. 2013;189(1 Suppl):S12-7; discussion S17. doi:10.1016/j.juro.2012.11.015
- 12. Minamida S, Satoh T, Tabata K, et al. Prevalence of fluoroquinolone-resistant Escherichia coli before and incidence of acute bacterial prostatitis after prostate biopsy. *Urology*. 2011;78(6):1235-1239. doi:10.1016/j.urology.2011.07.1392

- 13. Carlson WH, Bell DG, Lawen JG, Rendon RA. Multi-drug resistant E.coli urosepsis in physicians following transrectal ultrasound guided prostate biopsies--three cases including one death. *Can J Urol.* 2010;17(2):5135-5137.
- 14. Toren P, Razik R, Trachtenberg J. Catastrophic sepsis and hemorrhage following transrectal ultrasound guided prostate biopsies. *Can Urol Assoc J.* 2010;4(1):E12-4.
- 15. Al-Otaibi MF, Al-Taweel W, Bin-Saleh S, Herba M, Aprikian AG. Disseminated intravascular coagulation following transrectal ultrasound guided prostate biopsy. *J Urol.* 2004;171(1):346. doi:10.1097/01.ju.0000099351.37696.3a
- 16. Borer A, Gilad J, Sikuler E, Riesenberg K, Schlaeffer F, Buskila D. Fatal Clostridium sordellii ischio-rectal abscess with septicaemia complicating ultrasound-guided transrectal prostate biopsy. *J Infect*. 1999;38(2):128-129.
- 17. Erdogan H, Ekinci MN, Hoscan MB, Erdogan A, Arslan H. Acute bacterial meningitis after transrectal needle biopsy of the prostate: a case report. *Prostate Cancer Prostatic Dis.* 2008;11(2):207-208. doi:10.1038/pcan.2008.11
- 18. Dunfield L, Usman A, Fitzpatrick-Lewis D. Screening for prostate cancer with prostate specific antigen (PSA) and treatment of early-stage or screen-detected prostate cancer: a systematic review of the clinical benefits and harms. *Ottawa: Canadian Task Force on Preventive Health Care.* Published online 2013.
- 19. Venkatesan AM, Kundu S, Sacks D, et al. Practice guidelines for adult antibiotic prophylaxis during vascular and interventional radiology procedures. *J Vasc Interv Radiol*. 2010;21(11):1611-1630; quiz 1631. doi:10.1016/j.jvir.2010.07.018
- 20. Kubo Y, Kawakami S, Numao N, et al. Simple and effective local anesthesia for transperineal extended prostate biopsy: application to three-dimensional 26-core biopsy. *Int J Urol.* 2009;16(4):420-423. doi:10.1111/j.1442-2042.2009.02269.x
- 21. Meyer AR, Mamawala M, Winoker JS, et al. Transperineal Prostate Biopsy Improves the Detection of Clinically Significant Prostate Cancer among Men on Active Surveillance. *J Urol.* 2021;205(4):1069-1074. doi:10.1097/JU.000000000001523
- 22. Kasivisvanathan V, Dufour R, Moore CM, et al. Transperineal magnetic resonance image targeted prostate biopsy versus transperineal template prostate biopsy in the detection of clinically significant prostate cancer. *J Urol*. 2013;189(3):860-866. doi:10.1016/j.juro.2012.10.009
- 23. Radtke JP, Kuru TH, Boxler S, et al. Comparative analysis of transperineal template saturation prostate biopsy versus magnetic resonance imaging targeted biopsy with magnetic resonance imaging-ultrasound fusion guidance. *J Urol.* 2015;193(1):87-94. doi:10.1016/j.juro.2014.07.098

- 24. Huang H, Wang W, Lin T, et al. Comparison of the complications of traditional 12 cores transrectal prostate biopsy with image fusion guided transperineal prostate biopsy. *BMC Urol*. 2016;16(1):68. doi:10.1186/s12894-016-0185-z
- 25. Hansen NL, Kesch C, Barrett T, et al. Multicentre evaluation of targeted and systematic biopsies using magnetic resonance and ultrasound image-fusion guided transperineal prostate biopsy in patients with a previous negative biopsy. *BJU Int*. 2017;120(5):631638. doi:10.1111/bju.13711
- Siddiqui MM, Rais-Bahrami S, Turkbey B, et al. Comparison of MR/ultrasound fusionguided biopsy with ultrasound-guided biopsy for the diagnosis of prostate cancer. *JAMA*.
   2015;313(4):390-397. doi:10.1001/jama.2014.17942
- 27. Pokorny MR, de Rooij M, Duncan E, et al. Prospective study of diagnostic accuracy comparing prostate cancer detection by transrectal ultrasound-guided biopsy versus magnetic resonance (MR) imaging with subsequent MR-guided biopsy in men without previous prostate biopsies. *Eur Urol*. 2014;66(1):22-29. doi:10.1016/j.eururo.2014.03.002
- 28. Quentin M, Blondin D, Arsov C, et al. Prospective evaluation of magnetic resonance imaging guided in-bore prostate biopsy versus systematic transrectal ultrasound guided prostate biopsy in biopsy naïve men with elevated prostate specific antigen. *J Urol*. 2014;192(5):1374-1379. doi:10.1016/j.juro.2014.05.090
- 29. Arsov C, Rabenalt R, Blondin D, et al. Prospective randomized trial comparing magnetic resonance imaging (MRI)-guided in-bore biopsy to MRI-ultrasound fusion and transrectal ultrasound-guided prostate biopsy in patients with prior negative biopsies. *Eur Urol*. 2015;68(4):713-720. doi:10.1016/j.eururo.2015.06.008
- 30. Sonn GA, Margolis DJ, Marks LS. Target detection: magnetic resonance imagingultrasound fusion-guided prostate biopsy. *Urol Oncol.* 2014;32(6):903-911. doi:10.1016/j.urolonc.2013.08.006
- 31. Filson CP, Natarajan S, Margolis DJA, et al. Prostate cancer detection with magnetic resonance-ultrasound fusion biopsy: The role of systematic and targeted biopsies. *Cancer*. 2016;122(6):884-892. doi:10.1002/cncr.29874
- 32. Liu W, Patil D, Howard DH, et al. Impact of prebiopsy magnetic resonance imaging of the prostate on cancer detection and treatment patterns. *Urol Oncol*. 2019;37(3):181.e15-181.e21. doi:10.1016/j.urolonc.2018.11.004
- 33. Rosenkrantz AB, Hemingway J, Hughes DR, Duszak R, Allen B, Weinreb JC. Evolving use of prebiopsy prostate magnetic resonance imaging in the medicare population. *J Urol.* 2018;200(1):89-94. doi:10.1016/j.juro.2018.01.071
- 34. Bjurlin MA, Carroll PR, Eggener S, et al. Update of the standard operating procedure on the use of multiparametric magnetic resonance imaging for the diagnosis, staging and

management of prostate cancer. *J Urol.* 2020;203(4):706-712. doi:10.1097/JU.0000000000000017

- Meyer AR, Joice GA, Schwen ZR, Partin AW, Allaf ME, Gorin MA. Initial Experience Performing In-office Ultrasound-guided Transperineal Prostate Biopsy Under Local Anesthesia Using the PrecisionPoint Transperineal Access System. *Urology*. 2018;115:8-13. doi:10.1016/j.urology.2018.01.021
- 36. Perineologic, Allaway MJ. Perineologic. Accessed August 5, 2018. https://perineologic.com/
- 37. Liss MA, Ehdaie B, Loeb S, et al. An update of the American Urological Association white paper on the prevention and treatment of the more common complications related to prostate biopsy. *J Urol.* 2017;198(2):329-334. doi:10.1016/j.juro.2017.01.103
- 38. Urkmez A, Demirel C, Altok M, Bathala TK, Shapiro DD, Davis JW. Freehand versus Grid-Based Transperineal Prostate Biopsy: A Comparison of Anatomical Region Yield and Complications. *J Urol.* 2021;206(4):894-902. doi:10.1097/JU.000000000001902
- 39. Singer M, Deutschman CS, Seymour CW, et al. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). *JAMA*. 2016;315(8):801-810. doi:10.1001/jama.2016.0287
- 40. Zembower TR, Maxwell KM, Nadler RB, et al. Evaluation of targeted antimicrobial prophylaxis for transrectal ultrasound guided prostate biopsy: a prospective cohort trial. *BMC Infect Dis*. 2017;17(1):401. doi:10.1186/s12879-017-2470-1
- 41. Rosario DJ, Lane JA, Metcalfe C, et al. Short term outcomes of prostate biopsy in men tested for cancer by prostate specific antigen: prospective evaluation within ProtecT study. *BMJ*. 2012;344:d7894. doi:10.1136/bmj.d7894
- Lundström K-J, Drevin L, Carlsson S, et al. Nationwide population based study of infections after transrectal ultrasound guided prostate biopsy. *J Urol*. 2014;192(4):11161122. doi:10.1016/j.juro.2014.04.098
- 43. Bruyère F, Malavaud S, Bertrand P, et al. Prosbiotate: a multicenter, prospective analysis of infectious complications after prostate biopsy. *J Urol*. 2015;193(1):145-150. doi:10.1016/j.juro.2014.07.086
- 44. Wagenlehner FME, van Oostrum E, Tenke P, et al. Infective complications after prostate biopsy: outcome of the Global Prevalence Study of Infections in Urology (GPIU) 2010 and 2011, a prospective multinational multicentre prostate biopsy study. *Eur Urol*. 2013;63(3):521-527. doi:10.1016/j.eururo.2012.06.003
- 45. Loeb S, van den Heuvel S, Zhu X, Bangma CH, Schröder FH, Roobol MJ. Infectious complications and hospital admissions after prostate biopsy in a European randomized trial. *Eur Urol.* 2012;61(6):1110-1114. doi:10.1016/j.eururo.2011.12.058

- 46. Chambó RC, Tsuji FH, Yamamoto HA, Jesus CMN de. Short-term prophylaxis with ciprofloxacin in extended 16-core prostate biopsy. *Int Braz J Urol*. 2015;41(1):46-56. doi:10.1590/S1677-5538.IBJU.2015.01.08
- 47. Unnikrishnan R, El-Shafei A, Klein EA, Jones JS, Kartha G, Goldman HB. For single dosing, levofloxacin is superior to ciprofloxacin when combined with an aminoglycoside in preventing severe infections after prostate biopsy. *Urology*. 2015;85(6):1241-1246. doi:10.1016/j.urology.2014.12.062
- 48. Abughosh Z, Margolick J, Goldenberg SL, et al. A prospective randomized trial of povidone-iodine prophylactic cleansing of the rectum before transrectal ultrasound guided prostate biopsy. *J Urol.* 2013;189(4):1326-1331. doi:10.1016/j.juro.2012.09.121
- 49. Park DS, Hwang JH, Choi DK, et al. Control of infective complications of transrectal prostate biopsy. *Surg Infect (Larchmt)*. 2014;15(4):431-436. doi:10.1089/sur.2013.138
- 50. Ankerst DP, Straubinger J, Selig K, et al. A contemporary prostate biopsy risk calculator based on multiple heterogeneous cohorts. *Eur Urol*. 2018;74(2):197-203. doi:10.1016/j.eururo.2018.05.003
- 51. Lin DW, Newcomb LF, Brown MD, et al. Evaluating the Four Kallikrein Panel of the 4Kscore for Prediction of High-grade Prostate Cancer in Men in the Canary Prostate Active Surveillance Study. *Eur Urol.* 2017;72(3):448-454. doi:10.1016/j.eururo.2016.11.017
- 52. Vickers AJ, Elkin EB. Decision curve analysis: a novel method for evaluating prediction models. *Med Decis Making*. 2006;26(6):565-574. doi:10.1177/0272989X06295361

## **APPENDIX**

# Immediate post biopsy questionnaire

Please ask the patient to fill this out after the biopsy, before they leave the department.

Please check the box corresponding to the number, which describes how you felt immediately after the biopsy procedure:

1. Overall, how much **discomfort** did the biopsy procedure cause you? 4 5 7 9 10 3 No discomfort Moderate discomfort Extreme discomfort 2. Overall, how much pain did the biopsy procedure cause you? 4 8 9 10 1 2 3 5 6 No pain Moderate pain Extreme pain

3. Overall, how much **fear/anxiety** did the biopsy procedure cause you?

| | 0 | 1 | 2 | | 3 | 4 | 5 | 6 | | 7 | 8 | 9 | 10 | ) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | _ | | | | | | | | | | | |
| No fear or | anxiety | | | | ļ | Moder | ate fear o | r anxi | iety | | | Е | xtreme fe | ar or anxiety |
| 4 Plans | o list or | w mo | dica | tions t | that | . vou aro | currently | v tal | zina. | ۸n ov | amal | o ie giv | on in the | o firet |
| 4. Pleas box: | e iist ai | iy ille | uica | แบบร | ınaı | you are | currenti | y lar | King. | Allexa | ampi | e is giv | en in ui | z 1115t |
| ne of | | De | osag | ne er | | Numbe | | f | Star | t Date | | End [ | Date | Indicat |
| dication | | | | | ( | doses pe | er day | + | | | | | | |
| e.g. ciproflo | xacın | 5 | 00m | g | | 2 | | | 09/2 | 9/2021 | | 10/06/ | 2021 | Infection |
| | | | | | | | | + | | | | | | |
| Thank y | ou for | comi | olet | ina tl | he | auestio | nnaire. | Ple | ase | hand | this | to th | e resea | rch 7- |
| day pos | | | | | | | | | | | | | | |
| 1. Overa | all. how | much | dis | comf | ort | do vou h | nave fro | m th | e bio | psv? | | | | |
| | 0 | 1 | 2 | | 3 | 4 | 5 | 6 | | 7 | 8 | 9 | 10 | ) |
| No discom | fort | | | | | Mod | lerate disc | comfo | ort | | | | Extrem | e discomfort |
| 0 D | 1 | | - 4 41- | :4. | ! . | 41 1- | | 4. | - 1 ( | _ | | | | |
| 2. Do yo | ou nave | pain a | at tn<br>No | | wn | ere the b | iopsy w | as ta | aken | <b>?</b> | | | | |
| | l | | | | | | | | | | | | | |
| 3. If Yes | , how m | nuch <b>p</b> | ain | - | | having at | - | - | site? | | | | | |
| | 0 | 1 | 2 | | 3 | 4 | 5 | 6 | | 7 | 8 | 9 | 10 | ) |
| No pain | | | | I | | Mo | derate pai | n | | ı | | | E | Extreme pain |

| Dic | I you experience the following problems during the 7 days after the biopsy procedure? |
|---|---|
| 1. 1 | evers Yes No |
| 2.5 | Shivering and/or chills, as if you had a flu Yes No |
| 3.E | Blood in the urine ("pee" ) Yes No |
| 4.E | Blood in the semen (ejaculate or "cum" ) Yes No |
| 5. | Blood in the stools ("poop") Yes No |
| 6. | Acute urinary retention, meaning being unable to pass urine ("pee") which was relieved by putting a catheter into the bladder through the penis Yes No |
| 7. | Urinary tract infection diagnosed by a healthcare professional (doctor or nurse) Yes No |
| 8. | Please list any new medications, especially any painkillers or antibiotics, that you have taken since the biopsy. Do not list your regular medications but do list any new medications started related to the biopsy. Only list the medications if you have taken them. An example is given in the first box: Name of medication Dosage Number of doses per day Number of days |

| e.g. ciprofloxacin | 500mg | 2 | 3 |
|---|---|---|---|
| biopsy, which were unpl<br>Please answer yes if yo | anned and not<br>u have had any<br>ease also answe | s with hospital services for rea<br>part of the routine study visits?<br>unplanned contact with any he<br>er yes if you have had any unpl | ealthcare staff e.g. |
| unrelated to the biopsy? Please answer yes if yo e.g. GP, practice nurse, | u have had any<br>community nur | is with the community healthcare states, other. Please also answer ythcare staff over the phone: | aff in the community |

9.

| Thank you for questions. | completing | the question | naire. Please | contact us if | you have any |
|---|---|---|---|---|---|